CLINICAL TRIAL: NCT04638114
Title: Mini- Open Direct-anterior Approach vs Hip Arthroscopy for Treatment of Femoroacetabular Impingement. A Prospective Randomized Controlled Trial With 2 Years Follow up
Brief Title: Mini- Open Direct-anterior Approach vs Hip Arthroscopy for Treatment of Femoroacetabular Impingement.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator is no longer employed in study site
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: S53641
Record Dates: First submitted 2020-11-16; First posted 2020-11-20 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Femoracetabular Impingement
MeSH Terms: conditions — Femoracetabular Impingement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CAM lesion (Experimental): Mini-Open DAA Hip Arthroscopy
  Interventions: Procedure: Mini-open DAA; Procedure: Hip arthroscopy
- PINCER impingement (Other): Mini-Open DAA Hip Arthroscopy
  Interventions: Procedure: Mini-open DAA; Procedure: Hip arthroscopy

INTERVENTIONS:
Procedure: Mini-open DAA — Direct anterior approach hip
  Other Names: DAA
Procedure: Hip arthroscopy — arthroscopic treatment of hip pathology

SUMMARY:
Femoroacetabular impingement (FAI) is increasingly recognized as a common hip condition affecting the adolescent and adult population with groin pain and disability 1-5. When nonsteroidal anti-inflammatory medications, activity modification and injections fail as conservative treatment option fails, surgery addressing the underlying osseous pathoanatomy and associated labral and chondral lesions may be necessary.

Several techniques have been described as treatment of this condition. The first technique termed surgical hip dislocation (SHD) allowed to describe the pathomechanism of FAI 1, 3, 5, 6 and to develop treatment strategies such as osteochondroplasty, acetabular rim resection and fixation of torn labrum. Other techniques also have been proposed and consist of less invasive techniques as the (mini-open) direct anterior approach 7-10 and ´the golden standard´; the hip arthroscopy 11-15.

Good results have been reported for all techniques but faster rehabilitation and less morbidity have been published for hip arthroscopy (HA). The direct anterior approach also shows good results but a good randomized controlled trial to compare both techniques has not yet been performed.

Outcome is meanly determined by adequate bony correction of cam and pincer deformities. Direct visualization during SHD offers the advantage that possibly a more appropriate correction of the underlying morphology can be done. This thereby decreases the likelihood of early hip osteoarthritis (OA).

The purpose of the present study was to test the hypothesis that 1) the postoperative recovery and short term outcome after HA is superior compared to mini-open direct anterior approach and 2) the morphological corrections achieved by HA are equally sufficient when compared to the corrections achieved by the mini-open direct anterior technique.

DETAILED DESCRIPTION:
Hip arthroscopy versus mini-open direct anterior approach Surgical approach can have an important effect on post-operative recovery, complications and overall morbidity. Two frequently used approaches will be compared in the proposed study: the HA and the mini-open direct anterior approach. Outcome of HA vs mini-open direct anterior can thus be divided into clinical and morphological outcome parameters.

The clinical outcome parameters should be divided in early and long term outcome.

The early outcome is especially related to the surgery itself and postoperative rehabilitation. Outcome parameters are complication rate, hospital stay, blood loss, transfusion rate and functional recovery. The easiest way to describe functional outcome is by using internationally recognized and validated outcome scores. They are developed as an instrument to assess the patient's opinion about their hip and associated problems. These validated scores aim to assess the functionality and disability of the hip. The functional short and long term results of surgical procedures can be monitored with these outcome scores. In this study we use the Harris Hip Score, Hip disability and Osteoartritis Outcome Score (HOOS) and The Western Ontario and MacMaster (WOMAC) score. The Harris Hip Score (HHS) is probably one of the most frequently used scores to assess the outcome of procedures related to the hip joint16. Finally, the Hip disability and Osteoarthritis Outcome Score (HOOS) is a validated scoring system that consists of 39 items, divided into 5 sub-scales (i.e. pain, other symptoms, activity limitations in daily living (ADL), activity limitations in recreation and sport, and hip-related quality of life (QoL))17. The Western Ontario and MacMaster (WOMAC) is also a frequently used outcome tool and can be subtracted from the HOOS score18.

The late (>1 year) outcome parameters are the late complication rate and conversion to arthroplasty.

The morphological outcome is determined on anteroposterior pelvic x-rays and cross-table lateral views acquired preoperatively and 6 weeks after surgery. Several specific signs will be recorded. The presence of a cross-over sign 19 (COS), a posterior wall sign 19 (PWS), a prominence of the ischial spine 23 (PRISS) and a herniation pit 24 will be noted. Supplementary the CE-Angle 25, AC-Index 26, and quantitative COS 27 and the OA grade according to Tönnis 20 will be assessed. Additionally, the resection width angle 28 and the resection depth ratio 28 will be determined as schematically presented in Table 1.

On reconstructed radial reformations of arthro-CT scans acquired pre-operatively and 3 months after surgery, the alpha angle 18, anterior femoral head-neck offset 29, resection width angle, resection depth ratio, acetabular depth and the anterior acetabular coverage angle will be measured each on 7 positions from anterior to posterosuperior according to Locher 30 In summary, the proposed study is a randomized controlled study that focuses on the early and late clinical and morphological outcome parameters of the Hip Arthroscopy vs the mini-open direct anterior surgical approach in treatment of symptomatic femoroacetabular impingement.

Purpose of the study To assess surgical approach as a prognosticator for early and late functional recovery, complication rate and rate of morphological bony correction in patients with symptomatic femoroacetabular impingement Organisation This Randomised Controlled Trail (RCT) is set-up as a mono-center study. Surgeon: the prime investigator who will be perform all surgery . The patients will be pre-operatively randomly allocated (1:1 ratio) to either the HA or Mini-open direct anterior cohort.

Primary outcomes are formulated in terms of the Harris Hip Outcome score and morphological bony correction described by alpha angle, CE-angle and resection depth angle.

Secondary outcomes are the HOOS, WOMAC score, radiographic measures on AP pelvis view and arthro-CT as mentioned in Table 1 Contact with patients, surgery and follow-up will be done by the prime investigators but the functional and clinical assessments will be carried out by independent and blinded investigators trained in these investigations . These data will be prospectively collected in a protected database structure that allows for easy input and query assessment.

2. METHODS: PARTICIPANTS. All patients eligible for hip replacement surgery between August 2012 and December 2013 will be asked to participate the study in case they meet the inclusion criteria.

Inclusion criteria

Patients are eligible to be included when they meet the following criteria:

1. Age:

   - 15-80 years
2. Gender: 1:1 ratio of males and females / cohort
3. BMI: <30kg/m
4. Symptomatic FAI proven by clinical examination, plain radiographs and positive arthro-CT examination.
5. Clinical inclusion criteria: A positive impingement sign together with hip internal rotation in the 90° flexed hip position of less than 10° are the main clinical criteria.
6. Morphologic inclusion: a cam deformity (alpha angle higher 55°) 17 on radial arthro CT together with corresponding chondrolabral lesions

Exclusion criteria:

1. Previous surgery on their hip
2. Radiological investigations show acetabular retroversion with insufficient posterior wall (positive posterior wall sign) 19, additional acetabular dysplasia according to Lequesne's criteria 18, sequels of childhood hip disease such as Perthes disease or slipped capital femoral epiphysis, or hip OA higher to grade 1 according to Tönnis 20.
3. Neurologic impairment Reasons for withdrawal from the trial

1. Simple request by the patient, even without giving a reason. 2. Decision by the investigator, based upon suspicion of non-compliance by the patient.

3. Unexpected events not related to the surgical procedure such as serious illness that might impair the functionality of the patient.

Recruitment Recruitment will be done in the outpatient clinic. We reviewed a total of 26 patients who got a single- arthroscopic CAM resection in our centre by one single surgeon and measured a mean alpha-angle of 38° with a standard deviation of 7.5° after correction of the cam deformity. We assumed that if an alternative surgical technique would result in alpha angles differing less than 7.5° when compared to the angles after hip arthroscopy , this technique would be equivalent. Accordingly, a 7.5° difference was used for sample size calculation and revealed a number of 14 patients in each group in order to reject the null hypothesis with a significance level of 5% and a power of 80%.

We plan to include 20 patients in every group. This is certainly possible in a monocentric study.

Total minimum blinded follow-up is 2 years for the early outcomes and 5 and 10 years for the late outcome parameters.

Trial entry procedure The prime investigators will propose participation to the eligible patients in the outpatient clinic, as soon as surgery has been decided.

Patients will receive oral information and an 'Informed Consent form' with Patient information sheet' (see Addendum 1) for home study. This will give the patient time to think it over and to discuss it with the general practitioner, who will be informed by the investigator.

Randomisation will be done as soon as the patient agrees to join this trial. 3. METHODS: INTERVENTIONS General anaesthesia will be used for all surgeries. The arthroscopic technique, patient positioning and portal placements followed Byrd's 12 description using fluoroscopy. Osteochondroplasty will be intra-operatively with direct visualization an impingement-free flexion and internal rotation. The mini-open technique will be used as described by Clohisy 8.

For both techniques at least 30° of internal rotation in the 90° flexed hip position was the goal. Whereas weight bearing as tolerated on two crutches for 6 weeks was prescribed after HA, patients after mini-open technique will be prescribed touch weight bearing on two crutches as long as necessary for pain.

An independent and trained study nurse who will be blinded for the performed procedure will assess all patients at all time intervals. All patients will be assessed at the same time intervals: pre-operatively, 6w, 3-6-12-24months. The primary endpoints will already be assessed at a minimum follow-up of 12 months post-operatively as an intermediate and preliminary audit of the trial in order to detect any flaws and to re-evaluate the power-analysis.

4. METHODS: OBJECTIVES. To assess surgical approach as a prognosticator for early and late functional recovery, complication rate and rate of morphological bony correction in patients with symptomatic femoroacetabular impingement 5. METHODS: SAMPLE SIZE We reviewed a total of 26 patients who got a single- arthroscopic CAM resection in our centre by one single surgeon and measured a mean alpha-angle of 38° with a standard deviation of 7.5° after correction of the cam deformity. We assumed that if an alternative surgical technique would result in alpha angles differing less than 7.5° when compared to the angles after hip arthroscopy , this technique would be equivalent. Accordingly, a 7.5° difference was used for sample size calculation and revealed a number of 14 patients in each group in order to reject the null hypothesis with a significance level of 5% and a power of 80%.

We plan to include 20 patients in every group. This is certainly possible in a monocentric study.

Total minimum blinded follow-up is 2 years for the early outcomes and 5 and 10 years for the late outcome parameters.

6. METHODS: RANDOMIZATION. After the patient has agreed to joint trial and signed informed consent form, he or she will be assigned to the study and will be given a registration number.

This number will be signed on the sealed and non-transparent envelope that has been picked from the randomisation box. The envelope will be opened, the paper inside the envelope will first be signed with the registration number and the paper will then be unfolded.

The patient is then allocated to a study cohort and marked in the study database that is only accessible for the data monitor and the prime investigators.

Next the envelope is closed again and put into a sealed box until the end of the project.

The research nurse together with the patient will fill in the pre-operative clinical data.

7. METHODS: RANDOMIZATION. Randomisation will be done by 20 pieces of paper into a randomisation box signed with "HA" and 20 with "DAA". These pieces will be 4-folded so that the registration number of the patient can be written on the outside of the paper. The 40 pieces of paper will be put in sealed envelopes that are non-transparent and are put into one 'Randomisation box' by the data monitor.

The investigators will pick the envelope in the presence of the data monitor. A sealed 'Post-intervention box' will be created and all opened and signed envelopes and papers will be collected in this box that will only be accessible by the data monitor.

After patients have been assigned to a cohort they are scheduled for surgery. 8. METHODS: BLINDING (MASKING). Of course, the surgeon / prime investigator cannot be blinded. As a consequence he cannot be an assessor.

The patient will be blinded prior to surgery but will be able to differentiate the utilized approach based upon the incisions used.

The assessors however, namely the study nurse and evaluating junior-trainee will be blinded to the utilized approach. They will not be able to see the scar and the patient will be asked not to mention anything about the utilized approach. In case the patient would do this, than he or she will be excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 15-80 years
2. Gender: 1:1 ratio of males and females / cohort
3. BMI: <30kg/m
4. Symptomatic FAI proven by clinical examination, plain radiographs and positive arthro-CT examination.
5. Clinical inclusion criteria: A positive impingement sign together with hip internal rotation in the 90° flexed hip position of less than 10° are the main clinical criteria.
6. Morphologic inclusion: a cam deformity (alpha angle higher 55°) 17 on radial arthro CT together with corresponding chondrolabral lesions

Exclusion Criteria:

-

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-08; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Validated outcome score | 2 year
  Clinical outcome

SECONDARY OUTCOMES:
Radiographic measurement | 2 year
  Morphological Outcome parameter

CONTACTS AND LOCATIONS:
Overall Officials: Sigli Vanhooren, Study Chair
Locations (1):
- UZ Pellenberg, Pellenberg, Belgium

REFERENCES:
- [Result] Beck M, Leunig M, Parvizi J, Boutier V, Wyss D, Ganz R. Anterior femoroacetabular impingement: part II. Midterm results of surgical treatment. Clin Orthop Relat Res. 2004 Jan;(418):67-73. PMID 15043095